CLINICAL TRIAL: NCT06975124
Title: taVNS Effects on Fear Ratings in Naturalistic Context
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Weihua Zhao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UESTC-neuSCAN-100
Record Dates: First submitted 2025-04-23; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS group (Active Comparator): Eear clip electrodes were attached to the left cymba conchae to target vagus nerve branches.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Sham group (Sham Comparator): Electrode placements were attached on the left earlobe
  Interventions: Device: Sham condition

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Ear clip electrodes attached to the left cymba conchae to target vagus nerve branches.
  Arms: taVNS group
Device: Sham condition — Electrode placement attached on the left earlobe.
  Arms: Sham group

SUMMARY:
During the fear rating task, 70 participants viewed a 600-second horror movie while continuously rating their subjective fear intensity (0-100 scale) every 0.51 seconds (1,170 total ratings). Functional near-infrared spectroscopy (fNIRS) data were simultaneously recorded using the NIRSIT LITE system to monitor cortical hemodynamic responses.

DETAILED DESCRIPTION:
In a sham-controlled, participant-blinded, between-subjects design, 70 participants were randomly assigned to either active transcutaneous auricular vagus nerve stimulation (taVNS) or sham stimulation. The taVNS group received stimulation via a modified transcutaneous electrical acupoint stimulation device, with ear clip electrodes attached to the left cymba conchae to target vagus nerve branches. The sham group received identical electrode placement on the left earlobe, a non-vagus-innervated site. Stimulation intensity was individually calibrated to a perceptible but non-painful level to ensure vagal activation while maintaining participant comfort.

Upon arrival, all participants completed standardized mood and trait questionnaires. To assess emotional and physiological changes, two administrations of the Positive and Negative Affect Schedule (PANAS) and blood pressure/pulse measurements (pre- and post-intervention) were conducted. During the fear rating task, participants viewed a 600-second horror movie while continuously rating their subjective fear intensity (0-100 scale) every 0.51 seconds (1,170 total ratings). Functional near-infrared spectroscopy (fNIRS) data were simultaneously recorded using the NIRSIT LITE system to monitor cortical hemodynamic responses. Additionally, skin conductance responses were measured vy BIOPAC MP150 system.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants without color blindness, current or regular substance or medication use, any current or history of medical or psychiatric disorders and contraindications for MRI.

Exclusion Criteria:

* Color blindness,
* Current or regular substance or medication use
* any current or history of medical or psychiatric disorders and contraindications for MRI

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Neural activity changes between groups | 10 minutes
  The differences in the activity of frontal regions between groups using fNIRS
Fear ratings between groups | 10 minutes
  The differences in the fear ratings (0-100, from neutral to extremely fearful) between groups
Functional connectivity witnin frontal regions between groups | 10 minutes
  The differences in the functional connectivity within frontal regions using fNIRS between groups
The correlation between brain activity and behavioral ratings across groups | 10 minutes
  The correlation between brain activity and behavioral ratings across groups

SECONDARY OUTCOMES:
Skin conductance response between groups | 10 minutes
  The differences in the skin conductance response during watching video between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Nirsit Lite, Chengdu, Sichuan, China